CLINICAL TRIAL: NCT00525109
Title: Elevated Serum HDL in Four Generations of a Nashville Family
Status: Terminated | Type: Observational
Why Stopped: Unable to complete enrollment due lack of family interest.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, James Muldowney, Assistant Professor of Medicine, Vanderbilt University
Other Study IDs: 010535
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Hyperlipidemias
Keywords: Cholesterol; Hyperlipidemia; Gene array
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, Serum, DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Single family cohort
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No intervention

SUMMARY:
The purpose of this study is to determine the genetic basis of one family's hereditary hyper-HDL-emia using multiple modalities such as linkage analysis and gene array.

DETAILED DESCRIPTION:
HDL, or good cholesterol, has been shown to protect against heart attack and stroke. How HDL works as a protective agent is not well understood. There is a family that has 4 generations of living members with high HDL level. In the study, after consent is obtained, we will obtain 2 tablespoons of blood from all the family members in order to study their cholesterol levels and to obtain DNA in order to determine if there is a pattern of inheritance for this trait. We will also have them fill out a questionnaire about their medical history, diet and activity level as all of these can affect their HDL levels. In addition we will obtain additional blood (about 2 tablespoons) for plasma, white blood cells and also perform a biopsy to obtain skin cells from a matched pair of family members with and without the trait in order to determine which genes might be turned on and off because of this trait. We also wish to study other families who have members with high HDL cholesterol as well. These individuals will be identified from a core database.

ELIGIBILITY:
Inclusion Criteria:

* 26 living members of a family with HDL levels greater than 90mg/dl and several of whom will act as related age matched controls.
* The investigators will also identify individuals in a lipid core database with HDL's of greater than 90mg/dl who have normal or low LDL and triglyceride levels and determine if they have normal or low LDL and triglyceride levels and determine if they have family members (parents or siblings) who also have high HDL cholesterol.

Exclusion Criteria:

* Individuals who are not a member of the study family and individuals with high HDL's and elevated LDL and/or triglycerides.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Family
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2004-06; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas E Vaughan, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States